CLINICAL TRIAL: NCT07092293
Title: Using the Rehabilitation Treatment Specification System (RTSS) to Maximize Rehabilitation Research Impact: A Video-Based Observational Study
Brief Title: Studying Rehabilitation Treatments Using Video to Improve Recovery for Adults With Physical Disabilities
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Principal Investigator, Lauren Wengerd, Principal Investigator, Ohio State University
Other Study IDs: 2024H0351; GR138505 (Other Grant/Funding Number: American Occupational Therapy Foundation)
Record Dates: First submitted 2025-06-17; First posted 2025-07-29 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Spinal Cord Injury; Occupational Therapy
Keywords: occupational therapy; stroke; spinal cord injury
MeSH Terms: conditions — Stroke; Spinal Cord Injuries | interventions — Occupational Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Occupational Therapy Practitioners: Occupational therapists and occupational therapy assistants employed by OSU Wexner Medical Center
  Interventions: Other: occupational therapy
- Spinal Cord Injury: Spinal cord injury patients receiving outpatient OT at OSUMC
  Interventions: Other: occupational therapy
- Stroke: Stroke patients receiving outpatient OT at OSUMC
  Interventions: Other: occupational therapy

INTERVENTIONS:
Other: occupational therapy — N/A as there is no intervention for this study

SUMMARY:
This study aims to better understand how occupational therapists provide rehabilitation for adults recovering from stroke or spinal cord injury (SCI), with a focus on improving arm and hand function. Using video recordings of real outpatient therapy sessions, researchers will identify the key elements of treatment, such as the types of activities, the therapist's techniques, and how patients respond. The study will use the Rehabilitation Treatment Specification System (RTSS), a framework designed to clearly describe rehabilitation methods. By analyzing these sessions, the research team will develop a practical toolkit to help therapists and researchers deliver and study more effective rehabilitation treatments in the future.

ELIGIBILITY:
Occupational Therapy Inclusion Criteria:

* Must be a licensed OT practitioner (occupational therapist or occupational therapy assistant),
* The OT practitioner must treat at least one adult stroke or spinal cord injury patient with UE sensorimotor impairment per month
* The OT practitioner must be willing to be video recorded while treating their enrolled stroke or SCI patients.

Stroke Patients Inclusion Criteria:

* Must have a medical diagnosis of ischemic or hemorrhagic stroke
* Must be ≥ 18 years old
* Must have at least one OT goal related to UE hemiparesis
* Must have at least one remaining OT treatment session after enrollment
* The patient's OT must be enrolled in the study.

Spinal Cord Injury (SCI) Patients Inclusion Criteria:

* Must have a medical diagnosis of cervical spinal cord injury
* Must be ≥ 18 years old
* Must have at least one OT goal related to UE sensorimotor impairment
* Must have at least one remaining OT treatment session after enrollment
* The patient's OT must be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A purposive sample of OT practitioners working in an outpatient rehabilitation at OSUWMC will be recruited for this study.
  A purposive sample of stroke patients receiving OT at an OSU outpatient rehabilitation clinic will be recruited for this study.
  A purposive sample of SCI patients receiving OT at an OSU outpatient rehabilitation clinic will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time Spent on Different Types of Treatment Activities | Through study completion, Up to 24 months
  We will quantify time spent in different treatment types during standard care occupational therapy, as specified in the Rehabilitation Treatment Specification System.

SECONDARY OUTCOMES:
Feasibility of Video Recording Intervention | Following participant data collection/video recording through study completion, up to 24 months
  Feasibility of Intervention Measure - Participants will rate their acceptability of being video recorded through various questions on a 1-5 Likert scale where 1 is completely disagree and 5 is completely agree.
Acceptability of Video Recording Intervention | Following participant data collection/video recording through study completion, up to 24 months
  Acceptability of Intervention Measure (AIM) - Participants will gauge their acceptability and comfort with being video recorded. Participants will rate their acceptability of being video recorded through various questions on a 1-5 Likert scale where 1 is completely disagree and 5 is completely agree.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT07092293/Prot_SAP_000.pdf
  • Informed Consent Form: Patient Informed Consent Form (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT07092293/ICF_002.pdf
  • Informed Consent Form: OT Informed Consent Form (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT07092293/ICF_001.pdf